CLINICAL TRIAL: NCT06711562
Title: Model-informed Individualized Treatment of Anti-infective Drugs in Patients With Osteoarticular Infections
Brief Title: Model-informed Individualized Treatment of Anti-infective Drugs
Status: Recruiting | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: SDU-2024-BJ-005
Record Dates: First submitted 2024-10-28; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Osteoarticular Infections
MeSH Terms: interventions — Anti-Infective Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anti-Infective Drugs — Anti-infective drugs are administered using the traditional clinical dosing regimen, with no interventions.

SUMMARY:
The study aims to optimize individualized treatment of anti-infective drugs in osteoarticular infections by analyzing drug exposure in patients blood and/or tissues using population pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected/confirmed osteoarticular infections who are undergoing anti-infective drug therapy.

Exclusion Criteria:

* Pregnant/lactating women.
* There are other factors that the researchers think are not suitable for inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected/confirmed osteoarticular infections who are undergoing anti-infective drug therapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Clearance (L/h) | Through study completion, an average of 30 days
Volume of Distribution (L) | Through study completion, an average of 30 days

SECONDARY OUTCOMES:
ratio of the area under the concentration-time curve from 0 to 24 hours | Through study completion, an average of 30 days
  For time-dependent antimicrobials, the PD target is defined as the time of free drug concentration beyond MIC during the dose interval. For concentration-dependent antimicrobials, the PD target is defined as the ratio of the area under the concentration-time curve from 0 to 24 hours to the MIC.
erythrocyte sedimentation rate | Through study completion, an average of 30 days
  Clinical treatment outcome
Adverse events | Through study completion, an average of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Ph.D, Principal Investigator — Shandong University
Locations (1):
- Shandong Public Health Clinical Center, Jinan, China

IPD SHARING:
Plan to Share IPD: Undecided